CLINICAL TRIAL: NCT03970954
Title: Regulatory T-cell Induction by Low-dose Interleukin-2 in Women With Unexplained Repeated Spontaneous Early Miscarriages
Brief Title: Low-dose Interleukin-2 in Women With Unexplained Miscarriages
Acronym: FaCIL-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP180256
Record Dates: First submitted 2019-03-14; First posted 2019-06-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Miscarriage
Keywords: Low-dose Interleukin-2; Miscarriage; Regulatory T cells
MeSH Terms: conditions — Abortion, Habitual; Abortion, Spontaneous | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1 (Experimental): Low-dose IL-2
  Interventions: Drug: low-dose IL-2

INTERVENTIONS:
Drug: low-dose IL-2 — Subcutaneous injection of low dose of IL-2 for induction course of 5 days, the 10th day after the beginning of periods. At most 5 courses of low dose of IL-2.
  Other Names: interleukin-2

SUMMARY:
The purpose of this study is to demonstrate the ability of low dose IL-2 to stimulate peripheral blood Tregs of women with unexplained repeated early spontaneous miscarriages for development of a therapy to prevent fetal rejection by low dose IL-2.

DETAILED DESCRIPTION:
About 1 to 3% of women of childbearing age have repeated early spontaneous miscarriages that may be related to parental chromosomal abnormalities, uterine abnormalities, hormonal causes, infectious etiology, thrombophilia ... When one of these known causes is excluded, it is unexplained miscarriages of which half would be due to an immunological deregulation of the mother causing a decrease of the tolerance to the fetus.

In this context, the stimulation of regulatory T cells (Tregs) by low dose IL-2 is a therapeutic option with a rational, preclinical and clinical data very favorable.

In humans, low dose IL-2 allows preferential activation of Tregs and is very well tolerated. Several therapeutic trials have shown its efficiencies.

These elements make it possible to envisage the development of a therapeutic to prevent fetal rejection by IL2-fd on the women with spontaneous miscarriages by an immunological deregulation.

ELIGIBILITY:
Inclusion Criteria:

* Woman with at least 5 consecutive early miscarriages less than 14 weeks of amenorrhea and unexplained after the usual check-up;
* Volunteer to participate in the trial and having given written consent after appropriate information.

Exclusion Criteria:

* Uterine or pelvic abnormality: uterine malformation, intracavitary fibroid, synechiae, polyp, hydrosalpinx;
* Balanced translocations in both spouses;
* Diabetes type I or II;
* Sickle cell disease;
* Contraindication to pregnancy;
* Constitutional or acquired thrombophilia (protein deficit C, S, ATIII, homozygous factor V or II deficiency, antiphospholipid syndrome, antithyroid antibodies positive, celiac disease, hyperhomocysteinemia);
* Ovarian insufficiency (AMH <1 ng/ml); AFC < 4
* Significant spermogram abnormalities and DNA fragmented more than 30%
* Active HIV or HCV infection;
* Main known contraindications to treatment with IL-2:
* Hypersensitivity to the active substance or to any of the excipients;
* Signs of progressive infection requiring antibiotic therapy;
* History of organ allograft;
* Pre-existing autoimmune disease;
* Leukocytes <4000 / mm3; platelets <100,000 / mm3; hematocrit <30%;
* hepatic or renal insufficiency;
* depression;
* significant history or existence of a serious heart disease (in doubtful cases, perform a stress test);
* patients with autoimmune disease;
* patients with an infection (septicemia, bacterial endocarditis, septic thrombophlebitis, peritonitis and pneumonia);
* pregnancy;
* Treatment with immunomodulators, immunosuppressants (class L04A of the ATC classification), in particular systemic corticosteroids, as well as aspirin and low molecular weight heparin;
* No affiliation to a social security;
* Person who has already been included in this study or in another at the same time;
* Major incapacitated patient (tutorship / curatorship);
* Patient with an allergy to taking IL2-fd;
* Participants who would present professional risk factors (eg ionizing exposure);

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Variation of rate of blood circulating T regulator lymphocytes(expressed in % of CD4 and total) | At the day 38 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 1]
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2
Variation of rate of blood circulating T regulator lymphocytes(expressed in % of CD4 and total) | At the day 66 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 1
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2
Variation of rate of blood circulating T regulator lymphocytes(expressed in % of CD4 and total) | At the day 94 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 1
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2
Variation of rate of blood circulating T regulator lymphocytes(expressed in % of CD4 and total) | At the day 122 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 1
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2
Variation of rate of blood circulating T regulator lymphocytes(expressed in % of CD4 and total) | At the day 150 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 11
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2

SECONDARY OUTCOMES:
Variation of rate of blood circulating T regulator lymphocytes(expressed in absolute numbers) | At the day 38 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 1
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2
Variation of rate of blood circulating T regulator lymphocytes(expressed in absolute numbers) | At the day 66 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 1
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2
Variation of rate of blood circulating T regulator lymphocytes(expressed in absolute numbers) | At the day 94 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 1
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2
Variation of rate of blood circulating T regulator lymphocytes(expressed in absolute numbers) | At the day 122 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 1
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2
Variation of rate of blood circulating T regulator lymphocytes(expressed in absolute numbers) | At the day 150 of Cycle 2 (each cycle is 28 days) compared from the day 10 of Cycle 11
  Change of Tregs at Day 14 of cycles under low dose of IL-2 compared to the baseline of the first cycle without low dose of IL-2

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, Pr, Principal Investigator — Pitié Salpètrière APHP Paris; Arsene Mékinian, Dr, Study Director — Saint Antoine APHP Paris; Gilles Kayem, Pr, Study Director — Trousseau APHP Paris
Locations (3):
- France (3):
  - Mekinian, Paris, Hopital Saint Antoine
  - Bornes, Paris, Hopital Tenon
  - Kayem, Paris, Hopital Trousseau

IPD SHARING:
Plan to Share IPD: No